CLINICAL TRIAL: NCT04035824
Title: Evidence-based Optimization of Gastrodia and Uncaria Recipe in Treating Stage-one Hypertension: a Multi-center, Randomized, Double-blind, Placebo Controlled Trial
Brief Title: Gastrodia and Uncaria Recipe in Treating Stage-one Hypertension: an Evidence-based Optimization Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Institute of Hypertension (Other)
Collaborators: Ruijin Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yan Li, Professor, Vice Director of the Center for Epidemiological Studies and Clinical Trials, and Vice Director of the Center for Vascular Evaluations, Shanghai Institute of Hypertension
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018YFC1704902
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hypertension
Keywords: Gastrodia and Uncaria; Stage one Hypertension; Liver yang hyperactivity
MeSH Terms: conditions — Hypertension | interventions — gastrodin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gastrodia and Uncaria granule (Active Comparator): Gastrodia and Uncaria granule, Chengdu Jiuzhitang Jinding Pharmaceutical Co., Ltd
  Interventions: Drug: Gastrodia and Uncaria granule
- Placebo (Placebo Comparator): Placebo of Gastrodia and Uncaria granule, Chengdu Jiuzhitang Jinding Pharmaceutical Co., Ltd
  Interventions: Drug: Placebo of Gastrodia and Uncaria granule

INTERVENTIONS:
Drug: Gastrodia and Uncaria granule — Patients allocated to the intervention group take 10g of Gastrodia and Uncaria granule each time, twice per day, and for two months.
  Arms: Gastrodia and Uncaria granule
Drug: Placebo of Gastrodia and Uncaria granule — Patients allocated to the control group take 10g of placebo of Gastrodia and Uncaria granule each time, twice per day, and for two months. The placebo has similar appearance and smell to genuine drug but has no effective anti-hypertensive agents.
  Arms: Placebo

SUMMARY:
Gastrodia and Uncaria Recipe is a well-known effective prescription in Traditional Chinese Medicine (TCM) to treat hypertension of liver yang hyperactivity type, which manifests symptom of headache or dizziness. However, it lacks consolidated evidence by multi-center randomized controlled trials. The hypothesis of this study is that Gastrodia and Uncaria granule may have significant anti-hypertensive effect on patients with stage-one hypertension and liver-yang hyperactivity syndrome than placebo.

This study is a randomized, controlled, multi-center, double-blind clinical trial. This study aims to recruit 500 hypertension patients who 1) are untreated or taking anti-hypertensive medicine for at least two weeks and 2) have an office systolic blood pressure of 140-159 mmHg, an office diastolic blood pressure of <100 mmHg, and a 24-hour ambulatory mean systolic blood pressure of >=130 mmHg. The patients will be stratified according to center, sex, and the TCM type of liver yang hyperactivity/ liver yang non-hyperactivity, and are then randomly assigned to the treatment of Gastrodia and Uncaria granules or placebo for 2 months. The blood pressure lowering effect is evaluated by 24-hour ambulatory systolic blood pressure (primary outcome) / diastolic blood pressure, as well as by home and office blood pressures.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female sex, aged 18-80 years.
2. Not taking anti-hypertensive drugs for at least two weeks, or taking anti-hypertensive drugs for more than two weeks.
3. Office blood pressure averages of three consecutive readings per visit, at two screening visits all meet the limits: systolic blood pressure ranges from 140 to 159 mmHg, and diastolic blood pressure <100 mmHg.
4. 24h ambulatory mean systolic blood pressure >= 130mmHg.
5. Agreed to participant, able to join follow-up and to come to hospital at each visit.
6. Signed informed consent.

Exclusion Criteria:

1. Secondary hypertension, confirmed or suspected.
2. Failed at ambulatory blood pressure monitoring: effective reading < 70%, or the number of awakening BP reading <20, or sleep time BP reading <7.
3. Taking drugs that must be used for other diseases but have a potential effect on blood pressure, such as males taking alpha blockers for prostatic hypertrophy.
4. Having the onset of cardiovascular and cerebrovascular diseases such as stroke, myocardial infarction or heart failure within 6 months.
5. Having a history of atrial fibrillation or frequent arrhythmia.
6. Having abnormal lab test results: liver function (ALT, AST, TBL) ≥ 2 times the upper normal limit, or serum creatinine ≥ 176umol/L, or serum potassium ≥ 5.5mmol/L.
7. Pregnant or breastfeeding (for females).
8. Complicating other diseases that are not suitable for the trial, such as thyroid disease with active medication, acute infectious diseases, chronic mental illness, and tumors.
9. Possible poor compliance with the research process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory systolic blood pressure | 8 weeks
  The difference of change of 24h ambulatory systolic blood pressure after 8-week treatment between treatment and control group

SECONDARY OUTCOMES:
Change in office blood pressure | 4 and 8 weeks
  The difference of change of office systolic and diastolic blood pressure between treatment and control group
Change in 24-hour ambulatory systolic blood pressure by stratum | 8 weeks
  The difference of change of 24h ambulatory systolic blood pressure after 8-week treatment between liver yang hyperactivity and liver yang non-hyperactivity stratum
Change in 24-hour ambulatory diastolic blood pressure, daytime and nighttime blood pressure | 8 weeks
  The difference of blood pressure change of 24-hour mean ambulatory diastolic, daytime and nighttime systolic and diastolic between treatment and control group.
Change in home blood pressure | 8 weeks
  Difference of change of home systolic and diastolic blood pressure after 8-week treatment between treatment and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China